CLINICAL TRIAL: NCT02942290
Title: A Phase 1b Dose Escalation Study Evaluating the Safety and Pharmacokinetics of Venetoclax in Combination With Azacitidine in Subjects With Treatment-Naïve Higher-Risk Myelodysplastic Syndromes (MDS)
Brief Title: A Study Evaluating Venetoclax in Combination With Azacitidine in Participants With Treatment-Naïve Higher-Risk Myelodysplastic Syndromes (MDS)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M15-531; 2016-001657-41 (EudraCT Number); 2023-507154-32-00 (Other: EU CT)
Record Dates: First submitted 2016-10-18; First posted 2016-10-24 (Estimated); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Myelodysplastic Syndromes (MDS)
Keywords: Higher-Risk (HR) Myelodysplastic Syndromes (MDS); Pharmacokinetic; Venetoclax; Azacitidine; Acute Myelogenous Leukemia; Myelodysplastic Syndromes (MDS); Treatment-Naïve Higher-Risk
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — Azacitidine; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Venetoclax + Azacitidine (Experimental)
  Interventions: Drug: Azacitidine; Drug: Venetoclax

INTERVENTIONS:
Drug: Azacitidine — Powder for injection; taken subcutaneously (SC) or intravenous (IV); Administered on Days 1-7 of 28 days cycle or Days 1-5 of Week 1 & Days 1-2 of Week 2 of 28 day cycle.
Drug: Venetoclax — Oral; Tablet
  Other Names: ABT-199; GDC-0199; VENCLEXTA

SUMMARY:
This is a Phase 1b, open-label, non-randomized, multicenter, dose-finding study evaluating venetoclax in combination with azacitidine in participants with treatment-naïve higher-risk MDS comprising a dose-escalation portion and a safety expansion portion.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have documented diagnosis of untreated de novo MDS with:

  * International Prognostic Scoring System (IPSS) risk categories Int-2 or High (minimum IPSS overall score of 1.5) OR Revised IPSS (IPSS-R) categories intermediate, high or very high (score of > 3) and
  * Presence of less than 20% bone marrow blasts per bone marrow biopsy/aspirate.
* Eastern Cooperative Oncology Group (ECOG) performance score of less than or equal to 2.

Exclusion Criteria:

* Participant has received prior therapy for MDS. (Prior supportive care in form of transfusions or growth factors, etc., is not considered prior therapy).
* Participant has received prior therapy with a BCL-2 Homology 3 (BH3) mimetic.
* Participant has a diagnosis other than previously untreated de novo MDS (as defined in the protocol) including:

  * MDS with IPSS risk categories Low or Int-1 (overall IPSS score < 1.5)
  * Therapy-related MDS (t-MDS).
  * MDS evolving from a pre-existing myeloproliferative neoplasm (MPN).
  * MDS/MPN including chronic myelomonocytic leukemia (CMML), atypical chronic myeloid leukemia (CML), juvenile myelomonocytic leukemia (JMML) and unclassifiable MDS/MPN.
* Participant has received allogeneic Hematopoietic Stem Cell Transplantation (HSCT) or solid organ transplantation.
* Participant has received a live attenuated vaccine within 4 weeks prior to the first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Estimated)
Dates: Start 2017-01-12 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
AUCt for Azacitidine | Up to 32 days
  Area under the plasma concentration-time curve (AUC) from 0 to the time of the last measurable concentration (AUCt) for azacitidine.
Cmax of venetoclax | Up to 32 days
  Maximum plasma concentration (Cmax) of venetoclax.
AUCt for venetoclax | Up to 32 days
  Area under the plasma concentration-time curve (AUC) from 0 to the time of the last measurable concentration (AUCt) for venetoclax.
Tmax of venetoclax | Up to 32 days
  Time to Cmax (peak time, Tmax) of venetoclax.
AUC[0 to infinity] for azacitidine | Up to 32 days
  Area under the plasma concentration-time curve from Time 0 to infinite time.
Recommended Phase 2 dose (RPTD) and dosing schedule of venetoclax in combination with azacitidine | Measured from Day 1 until Day 28 per dose level.
  The RPTD of venetoclax [co-administered venetoclax and azacitidine] will be determined during the dose escalation phase of the study. RPTD will be determined using available safety and pharmacokinetics data [upon completion of the dose escalation phase].
Half-life (t[1/2]) for azacitidine | Up to 32 days
  Terminal elimination half-life (t[1/2]) for azacitidine.
Cmax for azacitidine | Up to 32 days
  Maximum plasma concentration (Cmax) of azacitidine.
AUC[0-24] for venetoclax | Up to 32 days
  AUC over a 24-hour dose interval (AUC[0-24]) for venetoclax.
Clearance (CL) for azacitidine | Up to 32 days
  Clearance is defined as the volume of plasma cleared of the drug per unit time.
Tmax for azacitidine | Up to 32 days
  Time to Cmax (peak time, Tmax) of azacitidine.
Complete Remission (CR) Rate | Measured from Cycle 1 Day 1 as long as the participant continues to benefit, or until the occurrence of unacceptable toxicity, death, exercise of investigator discretion, or withdrawal of consent, and for an anticipated maximum duration of 24 months.
  Complete remission rate will be defined as the proportion of participants who achieved a complete response per the International Working Group (IWG) 2006 criteria for Myelodysplastic Syndromes (MDS).

SECONDARY OUTCOMES:
Rate of red blood cell (RBC) transfusion independence | Measured from Cycle 1 Day 1 as long as the participant continues to benefit, or until the occurrence of unacceptable toxicity, death, exercise of investigator discretion, or withdrawal of consent, and for an anticipated maximum duration of 24 months.
  Percentages of participants who become RBC transfusion-independent.
Progression-Free Survival (PFS) | Measured from the date of first dose of study drug to the date of earliest disease progression or death due to disease progression or febrile neutropenia, and for an anticipated maximum duration of 24 months.
  PFS is defined as the number of days from the date of the first dose of study drug to the date of earliest disease progression or death due to disease progression or febrile neutropenia.
Overall Survival (OS) | Measured from the date of first dose of study drug to the date of death, and for up to 5 years after the last participant is enrolled.
  OS is defined as number of days from the date of first dose of the study drug to the date of death of any cause.
Hematologic Improvement (HI) rate | Measured from Cycle 1 Day 1 as long as the participant continues to benefit, or until the occurrence of unacceptable toxicity, death, exercise of investigator discretion, or withdrawal of consent, and for an anticipated maximum duration of 24 months.
  Percentages of participants with HI (erythroid/platelet/neutrophil responses).
Rate of platelet (PLT) transfusion independence | Measured from Cycle 1 Day 1 as long as the participant continues to benefit, or until the occurrence of unacceptable toxicity, death, exercise of investigator discretion, or withdrawal of consent, and for an anticipated maximum duration of 24 months.
  Percentages of participants who become platelet transfusion-independent.
Event-Free Survival (EFS) | Measured from the date of the first dose of study drug to the date of earliest disease progression, death of any cause and for up to 5 yrs after the last participant is enrolled
  Event-free survival (EFS) will be defined as the number of days from the date of the first dose of study drug to the date of earliest disease progression or death of any cause.
Time to transformation to acute myeloid leukemia (AML) | Measured from the date of first dose of study drug to date of documented AML transformation, defined as the presence of blast count greater than or equal to 20% in either peripheral blood or bone marrow for an anticipated maximum duration of 24 months.
  Defined as the number of days from the date of the first dose of study drug to the date of documented AML transformation.
Overall Response Rate (OR) | Measured from Cycle 1 Day 1 as long as the participant continues to benefit, or until the occurrence of unacceptable toxicity, death, exercise of investigator discretion, or withdrawal of consent and for an anticipated maximum duration of 24 months.
  OR (equals the rates of complete remission [CR] + partial remission [PR]) of venetoclax in combination with azacitidine.
Time to next treatment (TTNT) | Measured from the first dose of study drug to start of new non-protocol specified MDS therapy, and for up to 5 years after the last participant is enrolled.
  Time to next treatment (TTNT) will be defined as the time from the first dose of study drug to start of new non-protocol specified MDS therapy or death from any cause.
Marrow Complete Remission (mCR) Rate | Measured from Cycle 1 Day 1 as long as the participant continues to benefit, or until the occurrence of unacceptable toxicity, death, exercise of investigator discretion, or withdrawal of consent, and for an anticipated maximum duration of 24 months.
  Defined as the proportion of participants who achieved a marrow complete response with or without hematological improvement per the International Working Group (IWG) 2006 criteria for Myelodysplastic Syndromes.
Modified Overall Response Rate (mOR) | Measured from Cycle 1 Day 1 as long as the participant continues to benefit, or until the occurrence of unacceptable toxicity, death, exercise of investigator discretion, or withdrawal of consent and for an anticipated maximum duration of 24 months.
  mOR (equals CR + PR + mCR) of venetoclax in combination with azacitidine.
Duration of CR | Measured from Cycle 1 Day 1 as long as the participant continues to benefit, or until the occurrence of unacceptable toxicity, death, exercise of investigator discretion, or withdrawal of consent, and for an anticipated maximum duration of 24 months.
  Duration of CR will be defined as the number of days from the date of first response CR to the earliest documentation of progressive disease or death of any cause, whichever occurs earlier.
Duration of mOR | Measured from Cycle 1 Day 1 as long as the participant continues to benefit, or until the occurrence of unacceptable toxicity, death, exercise of investigator discretion, or withdrawal of consent and for an anticipated maximum duration of 24 months.
  Duration of response (mOR) will be defined as the number of days from the date of first response (CR, PR or mCR) to the earliest documentation of progressive disease or death of any cause, whichever occurs earlier.
Duration of OR | Measured from Cycle 1 Day 1 as long as the participant continues to benefit, or until the occurrence of unacceptable toxicity, death, exercise of investigator discretion, or withdrawal of consent and for an anticipated maximum duration of 24 months.
  Duration of response (OR) will be defined as the number of days from the date of first response (CR or PR) to the earliest documentation of progressive disease or death of any cause, whichever occurs earlier.
Rate of AML transformation | Measured from the date of first dose of study drug to date of documented AML transformation, defined as the presence of blast count greater than or equal to 20% in either peripheral blood or bone marrow for an anticipated maximum duration of 24 months.
  The AML transformation rate is defined as the proportion of participants transformed to Acute Myelogenous Leukemia.
Time to First Response (CR) | Measured from Cycle 1 Day 1 as long as the participant continues to benefit, or until the occurrence of unacceptable toxicity, death, exercise of investigator discretion, or withdrawal of consent, and for an anticipated maximum duration of 24 months.
  Time to first response (CR) will be defined as the number of days from the date of first dose of the study drug to the date of the first response of CR.
Time to First Response (mOR) | Measured from Cycle 1 Day 1 as long as the participant continues to benefit, or until the occurrence of unacceptable toxicity, death, exercise of investigator discretion, or withdrawal of consent and for an anticipated maximum duration of 24 months.
  Time to first response (mOR) will be defined as the number of days from the date of first dose of the study drug to the date of the first response of (CR, PR, or mCR).
Time to First Response (OR) | Measured from Cycle 1 Day 1 as long as the participant continues to benefit, or until the occurrence of unacceptable toxicity, death, exercise of investigator discretion, or withdrawal of consent and for an anticipated maximum duration of 24 months.
  Time to first response (OR) will be defined as the number of days from the date of first dose of the study drug to the date of the first response of (CR or PR).

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (37):
- United States (13):
  - Duplicate_University of Arizona Cancer Center - North Campus /ID# 154155, Tucson, Arizona
  - The University of Chicago Medical Center /ID# 153673, Chicago, Illinois
  - University of Maryland, Baltimore /ID# 153669, Baltimore, Maryland
  - Tufts Medical Center /ID# 153672, Boston, Massachusetts
  - Dana-Farber Cancer Institute /ID# 152735, Boston, Massachusetts
  - Washington University-School of Medicine /ID# 153671, St Louis, Missouri
  - Columbia University Medical Center /ID# 153661, New York, New York
  - Weill Cornell Medical College /ID# 155524, New York, New York
  - Oregon Medical Research Center /ID# 152734, Portland, Oregon
  - University of Pittsburgh MC /ID# 153662, Pittsburgh, Pennsylvania
  - Tennessee Oncology-Nashville Centennial /ID# 222769, Nashville, Tennessee
  - Vanderbilt University Medical Center /ID# 152738, Nashville, Tennessee
  - UT MD Anderson Cancer Center /ID# 153809, Houston, Texas
- Australia (9):
  - Concord Repatriation General Hospital /ID# 154958, Concord, New South Wales
  - Duplicate_St. Vincent's Hospital, Darlinghurst /ID# 222846, Darlinghurst, New South Wales
  - St George Hospital /ID# 154954, Kogarah, New South Wales
  - Liverpool Hospital /ID# 222410, Liverpool, New South Wales
  - Calvary Mater Newcastle /ID# 154957, Waratah, New South Wales
  - Duplicate_Princess Alexandra Hospital /ID# 154990, Woolloongabba, Queensland
  - Austin Health /ID# 154955, Heidelberg, Victoria
  - The Alfred Hospital /ID# 154956, Melbourne, Victoria
  - Fiona Stanley Hospital /ID# 222847, Murdoch, Western Australia
- Juravinski Cancer Centre /ID# 152947, Hamilton, Ontario, Canada
- France (2):
  - Centre Hospitalier Universitaire de Nantes, Hotel Dieu -HME /ID# 153828, Nantes, Pays de la Loire Region
  - Hôpital Saint-Louis /ID# 153827, Paris
- Germany (6):
  - Universitatsklinikum Mannheim /ID# 153140, Mannheim, Baden-Wurttemberg
  - Klinikum rechts der Isar /ID# 153139, Munich, Bavaria
  - Universitaetsklinikum Koeln /ID# 153141, Cologne, North Rhine-Westphalia
  - Duplicate_Universitaetsklinikum Carl Gus /ID# 153958, Dresden, Saxony
  - Universitaetsklinikum Leipzig /ID# 153142, Leipzig, Saxony
  - Universitaetsklinikum Halle (Saale) /ID# 153760, Halle
- Italy (2):
  - Duplicate_IRCCS AOU di Bologna - Policlinico Sant'Orsola-Malpighi /ID# 153763, Bologna, Emilia-Romagna
  - Duplicate_Azienda Ospedaliero-Universitaria Policlinico Umberto I /ID# 153764, Rome, Roma
- United Kingdom (4):
  - Norfolk and Norwich University Hospitals NHS Foundation Trust /ID# 156492, Norwich, Norfolk
  - Oxford University Hospitals NHS Foundation Trust /ID# 222567, Oxford, Oxfordshire
  - University Hospitals Birmingham NHS Foundation Trust /ID# 158810, Birmingham
  - King's College Hospital NHS Foundation Trust /ID# 156489, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garcia JS, Platzbecker U, Odenike O, Fleming S, Fong CY, Borate U, Jacoby MA, Nowak D, Baer MR, Peterlin P, Chyla B, Wang H, Ku G, Hoffman D, Potluri J, Garcia-Manero G. Efficacy and safety of venetoclax plus azacitidine for patients with treatment-naive high-risk myelodysplastic syndromes. Blood. 2025 Mar 13;145(11):1126-1135. doi: 10.1182/blood.2024025464. PMID 39652823
- See also: This clinical study may be evaluating a usage that is not currently FDA approved. Please see US Prescribing Information for approved uses. — http://rxabbvie.com/